CLINICAL TRIAL: NCT00541996
Title: A Randomized, Open-Label, Single-Dose, 4-Period Crossover, Comparative Bioavailability Study of 3 Sustained- Release Formulations and an Immediate- Release Formulation of Vabicaserin (SCA-136) in Healthy Subjects
Brief Title: Study Comparing Bioavailability of Oral Formulations of Vabicaserin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 3153A1-1116
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — vabicaserin

INTERVENTIONS:
Drug: vabicaserin

SUMMARY:
The purpose of this study is to determine the absorption rate of four oral formulations of vabicaserin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men aged 18-50 years.

Exclusion Criteria:

* Any significant disease state.
* History of drug or alcohol abuse within 1 year.
* Abnormal liver function tests.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-08; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Assess the bioavailability of four oral formulations of vabicaserin.

SECONDARY OUTCOMES:
Obtain additional safety and tolerability data for vabicaserin in healthy male subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Philadelphia, Pennsylvania, United States